CLINICAL TRIAL: NCT00835692
Title: A Relative Bioavailability Study of 500 mg Clarithromycin Tablets Under Fasting COnditions
Brief Title: Clarithromycin 500 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R02-663
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarithromycin Tablets (Experimental): Clarithromycin 500 mg Tablet (test) dosed in first period followed by Biaxin® 500 mg Tablet (reference) dosed in second period
  Interventions: Drug: Clarithromycin
- Biaxin® Tablets (Active Comparator): Biaxin® 500 mg Tablet (reference) dosed in first period followed by Clarithromycin 500 mg Tablet (test) dosed in second period
  Interventions: Drug: Biaxin®

INTERVENTIONS:
Drug: Clarithromycin — 500 mg Tablet
  Arms: Clarithromycin Tablets
Drug: Biaxin® — 500 mg Tablet
  Arms: Biaxin® Tablets

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 500 mg Clarithromycin Tablets with that of 500 mg BIAXIN® Tablets following a single oral dose (1 x 500 mg tablet) in healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

All subjects selected for this study will be healthy men or women 18 years of age or older at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.

Each subject will complete the screening process within 28 days prior to period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed and signed by each potential participant before full implementation of screening procedures.

Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.

The screening clinical laboratory procedures will include:

* HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
* CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
* HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens
* URINALYSIS: by dipstick; full microscopic examination if dipstick positive
* URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
* SERUM PREGNANCY SCREEN (female subjects only)
* FOLLICLE STIMULATING HORMONE (FSH; female subjects only): verify postmenopausal status

If female and :

is postmenopausal for at least 1 year; or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

Subjects with a recent history of drug or alcohol addiction or abuse. Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).

Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.

Subjects demonstration a positive hepatitis B surface antigen screen, hepatitis C antibody screen or a reactive HIV antibody screen.

Subjects demonstrating a positive drug abuse screen when screened for this study.

Female subjects who are currently breast feeding. Female subjects who are demonstrating a positive pregnancy screen. Subjects with a history of allergic response(s) to Clarithromycin or related drugs.

Subjects with a history of clinically significant allergies including drug allergies.

Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).

Subjects who currently use or reports using tobacco or nicotine-containing products within 90 days prior to Period I dosing.

Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.

Subjects who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will by advised not to donate blood for four weeks after completing the study.

Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.

Subjects who report receiving any investigational drug within 30 days prior to Period I dosing.

Subjects who report taking any prescription medication in the 14 days prior to Period I dosing, with the exception of topical products without systemic absorption.

Subjects who have been on an abnormal diet during the 28 days prior to Period I dosing.

Subjects who report an intolerance of direct venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS
Locations (2):
- United States (2):
  - PRACS Institute Ltd, East Grand Forks, Minnesota
  - PRACS Institute Ltd, Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Clarithromycin (Test) First: Clarithromycin 500 mg Tablet (test) dosed in first period followed by Biaxin® 500 mg Tablet (reference) dosed in second period
- Biaxin® (Reference) First: Biaxin® 500 mg Tablet (reference) dosed in first period followed by Clarithromycin 500 mg Tablet dosed in second period
Period: First Intervention
Arm/Group | Clarithromycin (Test) First | Biaxin® (Reference) First
Started | 28 | 28
Completed | 27 | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout
Arm/Group | Clarithromycin (Test) First | Biaxin® (Reference) First
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Clarithromycin (Test) First | Biaxin® (Reference) First
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clarithromycin (Test) First | Biaxin® (Reference) First | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 26 | 26 | 52
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 27 | 23 | 50
  Hispanic | 1 | 2 | 3
  Asian | 0 | 2 | 2
  Black | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Clarithromycin: Clarithromycin 500 mg Tablet (test) dosed in either period
- Biaxin®: Biaxin® 500 mg Tablet (reference) dosed in either period
Arm/Group | Clarithromycin | Biaxin®
Number analyzed (Participants) | 55 | 55
ng/mL | 2170.964 (690.215) | 2214.636 (763.844)
Statistical Analysis 1: Comparison: Clarithromycin vs Biaxin®; Test type: Non-Inferiority or Equivalence — The pharmacokinetic parameters will be evaluated statistically by an analysis of variance (ANOVA) appropriate for the experimental design of this study; Test/Ref Ratio of LS Mean x 100 = 98.4, 90% CI [91.5 to 106] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Clarithromycin | Biaxin®
Number analyzed (Participants) | 55 | 55
ng*h/mL | 17380.442 (6167.362) | 18481.089 (5728.638)
Statistical Analysis 1: Comparison: Clarithromycin vs Biaxin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 93.5, 90% CI [89.6 to 97.6] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Clarithromycin | Biaxin®
Number analyzed (Participants) | 55 | 55
ng*h/mL | 17265.639 (6136.361) | 18362.380 (5719.467)
Statistical Analysis 1: Comparison: Clarithromycin vs Biaxin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 93.5, 90% CI [89.5 to 97.7] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.